CLINICAL TRIAL: NCT04051125
Title: Evaluation of Anticholinergic Load Using the ACB "Anticholinergic Cognitive Burden" Scale in Parkinson's Patients
Brief Title: Evaluation of Anticholinergic Load
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0279
Record Dates: First submitted 2019-07-08; First posted 2019-08-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Drugs with anticholinergic properties may cause central and peripheral side effects. Several scales have been developed to evaluate the anticholinergic effect of drugs. Numerous studies have been published, showing a link between the anticholinergic load and the occurrence of adverse effects in the elderly.

Anticholinergic Cognitive Burden is a scale that identifies the severity of adverse effects of anticholinergic drugs specifically on cognition including cognitive decline, mental confusion, mild cognitive impairment, and dementia. It was developed from reviews of the medical literature and the calculation of drug affinities for muscarinic receptors. This list of drugs was presented to a team of experts including geriatricians, psychogeriatrists geriatric nurses and pharmacists, who assigned these drugs three scores ranging from 1 to 3:

* score 1: drugs with a possible anticholinergic effect on cognition demonstrated in vitro by its affinity for the muscarinic receptor or by calculation of the ASA level (anticholinergic activity of the serum), but without relevant clinical evidence of cognitive adverse effects;
* scores 2 and 3: drugs whose moderate or severe anticholinergic effect on cognition has been clearly established clinically. The drugs of scores 2 or 3 are differentiated by their ability to cause confusion and their properties to penetrate or not the blood-brain barrier.

The sum of the scores of the different drugs taken by the patient determines the cumulative cognitive risk score related to anticholinergics.

This ACB scale seems to be the most relevant in Parkinsonian patients.

Parkinson's disease (PD) is described for the first time in 1817 by an English doctor who gives it his name.

Parkinson's disease is a chronic, slowly progressive condition defined by the presence of motor symptoms (resting tremor, slowness and difficulty of movement or bradykinesia, muscle rigidity, equilibrium disorders) associated with variable non-motor symptoms ( such as constipation, fatigue, depression and anxiety, sleep disorders, impaired sense of smell, cognitive disorders). Age is the main risk factor for the disease (?).

There is a significant increase in the number of cases due to the aging of the population and the improvement in life expectancy.

By 2030, the number of Parkinson's patients could increase by 56% with 1 in 120 people over 45 with the disease.

Parkinsonian patients are subjected to a higher anticholinergic load, by the therapeutics used in their pathologies (antidepressants, neuroleptics, antiparkinsonians, etc ...).

These central and peripheral anticholinergic effects may add to the symptomatology in Parkinson's patients and aggravate their pathology.

My study project aims to improve the management of elderly patients with Parkinson's disease.

Hypothesis: People involved in the management of Parkinson's patients are not always aware of the potential anticholinergic effects of drugs. Indeed, anticholinergic effects can be responsible for many hospitalizations in the elderly.

This is why we want to make an inventory of treatments in Parkinson's patients at the entrance of hospitalization by evaluating the anticholinergic load using the ACB scale and the hospitalization exit in order to know if this score changed after informing the doctors responsible

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parkinson's patient
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of anticholinergic load | 1 day
  assessing the anticholinergic load using the scale ACB " Anticholinergic Cognitif Burden ". Anticholinergic Cognitive Burden is a scale to identify the severity of adverse effects of anticholinergic drugs specifically on cognition including cognitive decline, mental confusion, mild cognitive impairment, and dementia

CONTACTS AND LOCATIONS:
Overall Officials: FAURE DELINGER, DOCTOR, Study Director — UH MONTPELLIER
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC